CLINICAL TRIAL: NCT01356511
Title: High-dose Dexamethasone and Conventional Dose Prednisone, for the First-line Treatment of Adults With ITP: a Multicenter, Randomized Controlled, Clinical Trial
Brief Title: High-dose Dexamethasone Versus Conventional Dose Prednisone for Initial Treatment of Primary Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Peking Union Medical College Hospital (Other); Ruijin Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Tongji Hospital (Other); Shandong University of Traditional Chinese Medicine (Other); Anhui Provincial Hospital (Other Government); Zhejiang Provincial Hospital of TCM (Other); Second Hospital of Shanxi Medical University (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, Ming Hou, Prof, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-002
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2010-09

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
Keywords: Purpura, Thrombocytopenic, Idiopathic
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Prednisone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone group (Experimental): Patients in the PDN arm received PDNorally at 1.0mg/kg body weight daily for 4 consecutive weeks.
  Interventions: Drug: Prednisone
- Dexamethasone group (Experimental): DXM was administered orally at 40 mg daily for 4 consecutive days and then stopped
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Prednisone — Prednisone, po, 1 mg/kg/d, for 4 weeks.
  Other Names: CD-PRE
  Arms: Prednisone group
Drug: Dexamethasone — Dexamethasone, po, 40 mg/d, for 4 days.
  Other Names: HD-DXM
  Arms: Dexamethasone group

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University and other 11 well-known hospitals in China. In order to report the efficacy and safety of high-dose dexamethasone compared to conventional dose prednisone for the first-line treatment of adults with primary immune thrombocytopenia(ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicentre, randomised controlled trial of 300 adults with ITP from 11 medical centers in China. Part of the participants are randomly selected to receive high-dose dexamethasone treatment and the other part are selected to receive conventional dose of prednisone treatment. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. In order to report the efficacy and safety of high-dose dexamethasone compared to conventional dose prednisone for the first-line treatment of adults with ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. Untreated hospitalized patients, may be male or female, between the ages of 18 ~ 80 years.
3. To show a platelet count <30 * 10^9/L, and with bleeding manifestations.
4. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit.
3. Received high-dose steroids or IVIG in the 3 weeks prior to the start of the study.
4. Current HIV infection or hepatitis B virus or hepatitis C virus infections.
5. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
6. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.
7. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
8. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2010-09; Primary Completion 2014-05 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Proposed criteria for assessing response to ITP treatments | The time frame is up to 28 days per subject
  1. Complete response (CR)： A platelet count ≥ 100 * 10^9/L measured on two occasions > 7 days apart and the absence of bleeding.
  2. Response (R)： A platelet count ≥ 30 * 10^9/L and a greater than two fold increase in platelet count from baseline measured on two occasions > 7 days apart and the absence of bleeding.
  3. No response (NR)： A platelet count < 30 * 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, DR., Principal Investigator — Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Background] Cheng Y, Wong RS, Soo YO, Chui CH, Lau FY, Chan NP, Wong WS, Cheng G. Initial treatment of immune thrombocytopenic purpura with high-dose dexamethasone. N Engl J Med. 2003 Aug 28;349(9):831-6. doi: 10.1056/NEJMoa030254. PMID 12944568
- [Background] Mazzucconi MG, Fazi P, Bernasconi S, De Rossi G, Leone G, Gugliotta L, Vianelli N, Avvisati G, Rodeghiero F, Amendola A, Baronci C, Carbone C, Quattrin S, Fioritoni G, D'Alfonso G, Mandelli F; Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA) Thrombocytopenia Working Party. Therapy with high-dose dexamethasone (HD-DXM) in previously untreated patients affected by idiopathic thrombocytopenic purpura: a GIMEMA experience. Blood. 2007 Feb 15;109(4):1401-7. doi: 10.1182/blood-2005-12-015222. Epub 2006 Oct 31. PMID 17077333
- [Derived] Wei Y, Ji XB, Wang YW, Wang JX, Yang EQ, Wang ZC, Sang YQ, Bi ZM, Ren CA, Zhou F, Liu GQ, Peng J, Hou M. High-dose dexamethasone vs prednisone for treatment of adult immune thrombocytopenia: a prospective multicenter randomized trial. Blood. 2016 Jan 21;127(3):296-302; quiz 370. doi: 10.1182/blood-2015-07-659656. Epub 2015 Oct 19. PMID 26480931